CLINICAL TRIAL: NCT02366065
Title: Does Oral Acetaminophen Lower Intraocular Pressure?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Henry D. Jampel, M.D., M.H.S., Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIR00006973
Record Dates: First submitted 2015-01-28; First posted 2015-02-19 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acetaminophen (Experimental): study subjects will have their intraocular pressure measured at 8 am, 10 am, 12 pm and 4 pm. They will then take acetaminophen 650 mg qid for 7 days and the intraocular pressures again measured at 8 am, 10 am, 12 pm, and 4 pm. Subjects will then stop the acetaminophen and return one week later for one more set of intraocular pressure measurements at 8 am, 10 am, 12 pm, and 4 pm.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Before treatment, study subjects will have their intraocular pressure measured at 8 am, 10 am, 12 pm and 4 pm. They will then take acetaminophen 650 mg qid for 7 days and the intraocular pressures again measured at 8 am, 10 am, 12 pm, and 4 pm. Subjects will then stop the acetaminophen and return one week later for one more set of intraocular pressure measurements at 8 am, 10 am, 12 pm, and 4 pm.
  Other Names: tylenol

SUMMARY:
- Lowering intraocular pressure is the only proven treatment for glaucoma. Medications, almost always in the form of eye drops, are a mainstay for lowering intraocular pressure. Eye drops have the disadvantage of being difficult to administer and can have adverse effects on the surface of the eye and the surrounding tissues. Lowering intraocular pressure can be accomplished with oral carbonic anhydrase inhibitors, but the many systemic side effects of these agents relegates them to drugs of last resort. Therefore, an effective, well-tolerated, oral agent would be an important addition to the treatment of glaucoma. The hypothesis is that oral acetaminophen can lower intraocular pressure to a clinically significant degree in a dosing regimen that is both safe and convenient. The research is important because acetaminophen is inexpensive, available over-the-counter, and has a well known safety and side effect profile.

DETAILED DESCRIPTION:
* The study design is prospective case series. Before treatment, study subjects will have their intraocular pressure measured at 8 am, 10 am, 12 pm and 4 pm. They will then take acetaminophen 650 mg qid for 7 days and the intraocular pressures again measured at 8 am, 10 am, 12 pm, and 4 pm. Subjects will then stop the acetaminophen and return one week later for one more set of intraocular pressure measurements at 8 am, 10 am, 12 pm, and 4 pm. The subjects will receive a reminder, by phone or text message, the day before each visit. Although measurement of intraocular pressure is part of routine clinical care, multiple intraocular pressure measurements over the course of three different days is not.

  -- The subjects will not be masked to the intervention. The person measuring the intraocular pressure will be unaware of the purpose of the study, and hence there should be no bias in the measurement of the main outcome measure, intraocular pressure.
* Treatment will occur for 7 days only, and during that time we will not know if the treatment has been successful in lowering the intraocular pressure. The only basis upon which a participant would be removed would be if he or she reported adverse effects from the study medication before the one week.
* The rationale for choosing acetaminophen is that there are data that it may be effective in lowering intraocular pressure. The dose chosen for this study (650 mg qid), is a dosing regimen that is commonly used for the treatment of pain, and is below the maximum recommended daily dose of 3 gm/day. If this dosing scheme does NOT lower intraocular pressure, further investigations are not planned; if it does lower intraocular pressure, further studies will be performed to find the lowest effective dose.
* Acetaminophen has a several decades long safety record as an over the counter medication for the treatment of pain. The dose and route of administration proposed is standard. Many of the participants will likely have used acetaminophen in the past.

ELIGIBILITY:
Inclusion Criteria:

* not on intraocular pressure lowering medications for at least 6 weeks in either eye.
* IOP above 22 mm Hg and below 35 mm Hg in at least one eye. The eye with the higher IOP will be the study eye

Exclusion Criteria:

* using acetaminophen
* history of hepatic disease either reported by the patient or documented in the patient's medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lowering Eye Pressure | 7 days
  Eye pressure will be measured by using an IOP applanation tonometer seven days after the patient has stopped the medication.

CONTACTS AND LOCATIONS:
Overall Officials: Henry D Jampel, MD, Principal Investigator — Johns Hopkins University - Wilmer Eye Institute
Locations (1):
- Johns Hopkins - The Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Mohamed N, Meyer D. Intraocular pressure-lowering effect of oral paracetamol and its in vitro corneal penetration properties. Clin Ophthalmol. 2013;7:219-27. doi: 10.2147/OPTH.S38473. Epub 2013 Jan 30. PMID 23390358